CLINICAL TRIAL: NCT00098488
Title: A Phase 1 Study of 17-allylamino-17-demethoxygeldanamycin (17-AAG) (NSC 330507; IND 57,966) and Rituximab in Patients With Relapsed B-cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin With or Without Rituximab in Treating Patients With Relapsed B-Cell Chronic Lymphocytic Leukemia or Prolymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01460; OSU 0429; 2004C0058; NCI-6518; OSU-0429; CDR0000401516; R21CA115048 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Prolymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — tanespimycin; Rituximab

ARMS (1):
- Treatment (17-AGG and rituximab) (Experimental): Patients receive 17-AAG IV over 2 hours on days 1, 4, 8, 11, 15 and 18 (course 1). Patients achieving ≥ 25% reduction in measurable disease after course 1 receive an additional course of single-agent 17-AAG approximately 10 days later in the absence of disease progression or unacceptable toxicity and provided absolute lymphocyte count continues to decrease. Patients failing to achieve a 25% reduction in measurable disease after course 1 OR with disease progression after courses 1 or 2 of single-agent 17-AAG proceed to combination therapy comprising 17-AAG IV over 2 hours on days 1, 4, 8, 11, 15, 18, and 22; and rituximab IV over 4 hours on days 1 and 2 and over 1 hour on days 4, 8, 15, and 22 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tanespimycin; Biological: rituximab

INTERVENTIONS:
Drug: tanespimycin — Given IV
  Other Names: 17-AAG
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin when given with or without rituximab in treating patients with relapsed B-cell chronic lymphocytic leukemia or prolymphocytic leukemia. Drugs used in chemotherapy, such as 17-N-allylamino-17-demethoxygeldanamycin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Monoclonal antibodies may kill cancer cells that are left after chemotherapy. Giving 17-N-allylamino-17-demethoxygeldanamycin with or without rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of twice weekly 17-allylamino-17-demethoxygeldanamycin (17-AAG) in combination with weekly rituximab in patients with relapsed chronic lymphocytic leukemia (CLL).

II. To examine the pharmacology of twice weekly 17-AAG in combination with weekly rituximab in patients with relapsed CLL.

SECONDARY OBJECTIVES:

I. To evaluate toxicity (using NCI CTCAE v3.0 criteria) and preliminary efficacy of twice weekly 17-AAG when used in combination with weekly rituximab in this patient population.

II. To examine the kinetics of depletion of PDK1/AKT-related proteins, mutant p53 and up-regulation of alternative targets that mediate resistance to therapy following treatment with twice weekly 17-AAG; and the relationship of this to spontaneous and drug-induced apoptosis in patients with relapsed CLL.

III. To examine the immunologic effects of twice weekly 17-AAG, in conjunction with weekly rituximab, in patients with relapsed CLL.

IV. To evaluate toxicity and preliminary efficacy of twice weekly 17-AAG as a single agent in this patient population.

OUTLINE: This is a multicenter, dose-escalation study of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG).

Patients receive 17-AAG intravenously (IV) over 2 hours on days 1, 4, 8, 11, 15 and 18 (course 1). Patients achieving ≥ 25% reduction in measurable disease after course 1 receive an additional course of single-agent 17-AAG approximately 10 days later in the absence of disease progression or unacceptable toxicity and provided absolute lymphocyte count continues to decrease. Patients failing to achieve a 25% reduction in measurable disease after course 1 OR with disease progression after courses 1 or 2 of single-agent 17-AAG proceed to combination therapy comprising 17-AAG IV over 2 hours on days 1, 4, 8, 11, 15, 18, and 22; and rituximab IV over 4 hours on days 1 and 2 and over 1 hour on days 4, 8, 15, and 22 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of 17-AAG as a single agent or in combination with rituximab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed up at 2 months and then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed B-cell chronic lymphocytic leukemia or prolymphocytic leukemia requiring treatment, defined by 1 of the following criteria:

  * Massive or progressive splenomegaly and/or lymphadenopathy
  * Anemia (hemoglobin < 11 g/dL) OR thrombocytopenia (platelet count < 100,000/mm^3)
  * Weight loss > 10% within the past 6 months
  * Grade 2 or 3 fatigue
  * Fevers > 100.5°F or night sweats for > 2 weeks with no evidence of infection
  * Progressive lymphocytosis with an increase of > 50% over a 2 month period OR an anticipated doubling time of < 6 months
* Relapsed disease
* Failed prior fludarabine or pentostatin therapy OR cannot receive fludarabine
* Lymphocyte count ≥ 5,000/mm^3
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* Bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL
* LVEF > 40% by MUGA
* QTc < 450 msec for male patients and < 470 msec for female patients
* Resting ejection fraction ≥ 50% by MUGA or echocardiogram
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No significant cardiac disease including any of the following:

  * New York Heart Association class III or IV heart failure
  * History of myocardial infarction within the past year
  * History of uncontrolled dysrhythmias
  * Active ischemic heart disease within the past year
  * Poorly controlled angina
* No history of serious ventricular arrhythmia (e.g., ventricular fibrillation, history of symptomatic or sustained ventricular tachycardia, nonsustained ventricular tachycardia > 3 beats within the past 6 months)
* No history of cardiac toxicity due to anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, or mitoxantrone hydrochloride)
* No other cardiac symptoms ≥ grade 2
* DLCO (i.e., oxygen diffusion capacity) ≥ 80% by pulmonary function testing
* Resting and exercise oxygen saturation ≥ 90% by pulse oximetry
* No pulmonary symptoms ≥ grade 2
* No history of pulmonary toxicity due to bleomycin or carmustine
* No significant, symptomatic pulmonary disease requiring oxygen or medications
* No ongoing pulmonary symptoms ≥ grade 2 including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Significant pulmonary disease (e.g., chronic obstructive or restrictive pulmonary disease)
* No Medicare requirements for home oxygen (e.g., resting O_2 saturations ≥ 90% or desaturation to ≥ 90% with exertion)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to 17-N-allylamino-17-demethoxygeldanamycin
* No history of serious allergic reaction to eggs
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness that would preclude study participation
* More than 3 months since prior rituximab and recovered
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy that potentially included the heart in the field (e.g., mantle)
* No history of chest radiation
* No concurrent medications that prolong or may prolong QTc
* No concurrent antiarrhythmic drugs
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-04; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) | Week 4
  Defined at the dose level of 17-AAG at which 2 (or more) of 6 patients develop dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Minimally effective pharmacological dose (MEPD) of 17-AAG based on down-modulation of the target protein Akt | Day 1
  Defined as the 17-AAG dose achieving >= 50% reduction in Akt protein expression.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lin, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States